CLINICAL TRIAL: NCT00143845
Title: Phase II Trial of Adjuvant Cellular Immunotherapy for High-Risk Hematologic Malignancy After Reduced Intensity Allogeneic Stem Cell Transplantation
Brief Title: Study of Low-Intensity Conditioning for Allogeneic Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2-61
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Results first posted 2014-06-20 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Multiple Myeloma; Lymphocytic Leukemia, Chronic; Lymphoma, Low-Grade
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immunosuppression Taper (Experimental): Reduced intensity conditioning consisting of Busulfan and Fludarabine(fludarabine 150 mg/m2 IV, busulfan 6 mg/kg IV, total lymphoid irradiation 2 Gy), followed by a rapid immunosuppressive taper of Tacrolimus (0.06 mg/kg q12h, PO, Days -7 to +28), Methotrexate (5 mg/m2, IV, Days +1, +3, +6, +11) and Mycophenolate Mofetil (10 mg/kg every 8 hours, PO, Days -6 to +7).
  Interventions: Procedure: Reduced intensity conditioning; Procedure: Rapid immunosuppressive taper; Procedure: Prophylactic donor leukocyte infusions

INTERVENTIONS:
Procedure: Reduced intensity conditioning — Busulfan and Fludarabine regimen
Procedure: Rapid immunosuppressive taper — Taper of Tacrolimus, Methotrexate and Mycophenolate Mofetil
Procedure: Prophylactic donor leukocyte infusions — If the patient has GVHD overall grade 0-1 or skin grade 1 on day +100, then 5 x 107 CD3+ cells/kg recipient weight are given.

SUMMARY:
The purpose of this study is to determine whether a reduced intensity conditioning regimen for stem cell transplant with donor cells will allow the donor cells to be effective without causing health problems.

DETAILED DESCRIPTION:
In this research study patients will receive dosages of chemotherapy that are lower than the usual dosages. The study will determine whether a shorter duration of immunosuppression will permit the donor cells to be effective against the cancer without causing more severe GVHD (Graft Versus Host Disease). Also to be determined is whether the patient's cancer can be prevented from relapsing after blood stem cell transplant by using prophylactic treatment, giving a donor leukocyte infusion BEFORE a relapse happens.

In this research study samples of blood and bone marrow will be analyzed. These samples will be examined to study the cellular production of inflammatory cytokine levels in attempt to be able to predict which patients will have complications like GVHD or relapse.

ELIGIBILITY:
Patient Inclusion Criteria:

To be eligible a patient MUST meet at least one of the next 4 criteria

* Any patient aged 55 years or older with a hematological malignancy for which allogeneic transplant is considered an appropriate treatment, AND/OR
* Any patient, regardless of age, with a hematologic malignancy for which allogeneic transplant is considered an appropriate treatment and the patient is not eligible for a conventional myeloablative transplant because of organ dysfunction AND/OR
* Any patient, regardless of age, who has relapsed following prior autologous or allogeneic transplant for a hematologic malignancy AND/OR
* Any patient, regardless of age, with one of the following hematological malignancies:

  1. Multiple myeloma

     1. refractory to or failure following conventional chemotherapy such as VAD (Vincristine, Adriamycin and Dexamethasone), pulse decadron, or alkylating agents, or
     2. chromosomal abnormality associated with poor prognosis by cytogenetics or FISH probe.
  2. Chronic lymphocytic leukemia patients, Rai stage 3 or 4 and relapsed following/refractory to alkylating agents or nucleoside analog therapy
  3. Low grade lymphoma (small lymphocytic, follicular small cleaved cell, or follicular mixed small cleaved and large cell) that is either relapsed or refractory provided the disease is NOT rapidly progressive, NOT bulky, and no mass exceeds 5 cm in greatest dimension.

To be eligible a patient MUST meet all of the following criteria

* In addition to the above criteria ALL patients must meet the following minimum organ function:

  1. Cardiac: Ejection fraction at least 30%.
  2. Renal: Adequate renal function as defined by creatinine < 2.0mg OR creatinine clearance >40 mg/min by 24-hour urine collection or GFR (Glomerular Filtration Rate. (Gender and age-adjusted creatinine clearance >40ml/min by Gault-Cockroft 55 is acceptable for adults: (140 - age) x weight/72 x Scr [x 0.85 if female]).
  3. Pulmonary: FEV1 and FVC >60%.
  4. Hepatic: Total bilirubin <2.0 and AST (Aspartate Aminotransferase)/ALT (Alanine Transaminase) < 3X institutional normal for age.
  5. Performance (adults): Karnofsky score must be at least 60; for pts. under 16, Lansky score must be at least 60.
* Availability of a 5/6 or 6/6 HLA A, B, and DR identical relative who is willing and able to donate allogeneic stem cells. Serological, low resolution or mid resolution molecular typing will determine the degree of match for HLA (Human Leukocyte Antigen) class I regardless of high resolution DNA typing results. High resolution typing will be used to determine the degree of match for HLA-DR.
* No untreated or uncontrolled invasive infections. Patients still under therapy for presumed or proven infection are eligible provided there is clear evidence (radiologic and/or culture) that the infection is well controlled. Patients under treatment for infection will be enrolled only after clearance from the Principal Investigator.
* Not pregnant

Patient Exclusion Criteria:

* acute leukemia
* HIV positive patients not eligible
* Any physical or psychological condition that, in the opinion of the investigator, would pose unacceptable risk to the patient
* Pregnant

Donor Inclusion Criteria:

* 5/6 or 6/6 HLA match for HLA-A, B, and DR
* Age 3-70 years, good general health
* No contraindication to G-CSF (Granulocyte Colony-Stimulating Factor)stimulation
* No contraindication to leukapheresis of peripheral blood stem cells
* Good general health

Donor Exclusion Criteria:

* HIV positive or history of HIV risk factors
* Presence of other diseases transmissible by blood that pose unacceptable risk to the study subject.
* Pregnant
* Medical or psychological conditions that would make the donor unlikely to tolerate G-CSF - injections or leukapheresis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-04; Primary Completion 2010-11 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Levine, MD, MS, Principal Investigator — The Univeristy of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immunosuppression Taper
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 54 patients were enrolled however 9 patients did not receive planned donor lymphocyte infusion. 45 patients were analyzed.
Arm/Group | Immunosuppression Taper
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 56 [2 to 67]
Gender [Count of Participants; unit: Participants]
  Female | 22
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Acute Graft Versus Host Disease (GVHD) Grades 2-4
Description: The primary objective of this study was to establish the rate of acute GVHD following prophylactic cellular immunotherapy after allogeneic hematopoietic stem cell therapy using low intensity conditioning for high-risk hematological malignancies. Glucksberg staging was used for organ grading of GVHD. Clinical GVHD was assessed as follows:
  Grade 0: No stage 1-4 of any organ Grade 1: Stage 1-2 rash and no liver or gut involvement Grade 2: Stage 3 rash, or Stage 1 liver involvement, or Stage 1 GI Grade 3: Stage 0-3 skin with Stage 2-3 liver, or Stage 2-4 GI Grade 4: Stage 4 skin rash, or Stage 4 liver involvement
Time Frame: 100 days
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Immunosuppression Taper
Number analyzed (Participants) | 45
percentage of participants | 73

2. Primary Outcome: Percentage of Participants With Progression Free Survival
Description: The second primary objective was to determine the percentage of participants with progression free survival following prophylactic cellular immunotherapy after allogeneic hematopoietic stem cell therapy using low intensity conditioning for high-risk hematological malignancies.
  We define disease progression as disease recurrence within 180 days of transplant.
Time Frame: two years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Immunosuppression Taper
Number analyzed (Participants) | 45
percentage of participants | 35

3. Secondary Outcome: Percentage of Patients Alive at 2 Years
Description: To estimate the overall survival of patients progression following prophylactic cellular immunotherapy after allogeneic hematopoietic stem cell therapy using low intensity conditioning for high-risk hematological malignancies.
Time Frame: 2 Years
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Immunosuppression Taper
Number analyzed (Participants) | 45
percentage of participants | 38

ADVERSE EVENTS:
Arm/Group | Immunosuppression Taper
Serious Adverse Events (participants affected / at risk) | 42/54
Other Adverse Events (participants affected / at risk) | 30/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immunosuppression Taper (N=54)
Diarrhea (Gastrointestinal disorders) | 10
GVHD (Immune system disorders) | 9
DVT (Vascular disorders) | 1
Infection (Infections and infestations) | 16
Primary Graft Failure (General disorders) | 1
Fever (General disorders) | 5
Relapsed Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypotension (Cardiac disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Vertigo (Ear and labyrinth disorders) | 1
Headache (Nervous system disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Weakness (General disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Pyrexia (General disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Lipase (Investigations) | 1
Amylase (Investigations) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Supraventricular tachycardia (Cardiac disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Supraventricular arrhythmia (Cardiac disorders) | 1
GVHD with infectious complications (Immune system disorders) | 1
Death (General disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immunosuppression Taper (N=54)
Hypomagnesemia (Metabolism and nutrition disorders) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 29
Hypoglycemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 28
Hypercalcemia (Metabolism and nutrition disorders) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 16
Hyperkalemia (Metabolism and nutrition disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 17
Hyponatremia (Metabolism and nutrition disorders) | 20
Hypernatremia (Metabolism and nutrition disorders) | 5
Creatinine (Investigations) | 18
Esophogitis (Gastrointestinal disorders) | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 24
AST (Investigations) | 20
ALT (Investigations) | 20
ALK (Investigations) | 15
Rash (Skin and subcutaneous tissue disorders) | 5
Infection (Infections and infestations) | 10
Total Bilirubin (Investigations) | 10
Mucositis (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes